CLINICAL TRIAL: NCT06406387
Title: Association Between Endoscopic Ultrasound Based Preoperative ATRX/DAXX Immunohistochemistry Expression and Prognosis of Sporadic, Non-FunctiOnal pancREatic Neuroendocrine tumorS: a prospEctivE Cohort Study
Brief Title: ATRX/DAXX in EUS-FNB Specimens of Pan-NETs
Acronym: FORESEE
Status: Active, not recruiting | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Other Study IDs: FORESEE
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Neuroendocrine Tumor
MeSH Terms: conditions — Adenoma, Islet Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ATRX/DAXX loss: The "positive" group including patients with loss of DAXX or ATRX expression evaluated on immunohistochemistry on endoscopic ultrasound biopsy specimens
  Interventions: Diagnostic Test: ATRX/DAXX immunohistochemistry
- ATRX/DAXX preserved: The "negative" group including those with preserved DAXX and ATRX expression evaluated on immunohistochemistry on endoscopic ultrasound biopsy specimens
  Interventions: Diagnostic Test: ATRX/DAXX immunohistochemistry

INTERVENTIONS:
Diagnostic Test: ATRX/DAXX immunohistochemistry — Immunohistochemistry will be performed using an Autostainer Leica (Leica Biosystems) according to the manufacturer's instructions. Four μm formalin-fixed paraffin-embedded sections will be immunostained with antibodies for Cytokeratin AE1/AE3 (AE1-AE3, 1:100 dilution, Novocastra/United Kingdom) Chromogranin A (DAK-A3, 1:2500, Dako/Denmark), and Synaptophysin (27G12, 1:100, Novocastra), Ki67 (MIB1, 1:100, Dako/Denmark), ATRX (1:400, Sigma-Aldrich), DAXX (1:200, Sigma-Aldrich). After antigen retrieval, immunostaining will be performed in an automated Bond instrument (Vision-Biosystem, Leica, Milan, Italy) using a sensitive peroxidase-based 'Bond polymer Refine' detection system.

SUMMARY:
P-NENs are classified as functional (F-) or non-functional (NF-) depending on the presence or absence of a clinical hormonal hypersecretion syndrome. Moreover, the WHO 2017 classification of pNENs distinguishes between well-differentiated pancreatic neuroendocrine tumors (pNETs) and poorly differentiated pancreatic neuroendocrine carcinomas (pNECs). pNETs are then divided according to a grading scheme based on Ki67 index in pNETs-G1 (Ki67 index ≤3%) and pNETs-G2 (Ki67 index between 4% and 20%). pNECs are all G3, with a Ki67 index >20%. Endoscopic ultrasound with fine-needle biopsy (EUS-FNB) demonstrated safe and effective preoperative grading based on the Ki-67 proliferative index. However, downstaging rate is not neglectable, reaching 15% in a recent metanalysis. Moreover, recent whole-exome and whole genome sequencing studies revealed that the mutually exclusive inactivating mutations in death domain-associated protein (DAXX) and/or in α-thalassemia/mental retardation X-linked (ATRX) chromatin remodeling genes are associated with more aggressive disease. In a retrospective study, the investigators recently evaluated the correspondence of DAXX/ATRX expression on 41 EUS-FNB samples with corresponding surgical specimens demonstrating a 95.1% (almost perfect agreement, κ = 0.828; p < 0.001) and 92.7% (substantial agreement, κ = 0.626; p < 0.001) concordance for DAXX and ATRX expression, respectively. This study aims to evaluate the potential clinical/prognostic role of DAXX/ATRX expression as implementation of the currently used Ki67-based grading, evaluated on EUS-FNB samples in a prospective cohort of patients with NF-pNETs

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Cyto/histologic diagnosis of pNETs
* Signed informed consent

Exclusion Criteria:

* Functional pNETs
* Multiple pancreatic nodules
* Diagnosis of MEN-1 or Von-Hippel Lindau
* Mixed types (e.g., mixed neuroendocrine-acinar/adenocarcinoma) or neuroendocrine carcinomas
* Predominantly cystic lesions (more than 50% of the volume).
* Metastatic tumors at the time of diagnosis
* Known bleeding disorder that cannot be sufficiently corrected with co-fact or fresh frozen plasma
* Use of anticoagulants that cannot be discontinued
* INR >1.5 or platelet count <50.000
* Pregnancy or breastfeeding
* Failure to sign the patient's or closest relative's informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of pancreatic neuroendocrine tumors
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
ATRX/DAXX loss-tumor aggressiveness association | 18 months
  To assess the association between ATRX/DAXX loss of expression assessed on endoscopic ultrasound biopsy specimens and pathological features indicative of tumor aggressiveness evaluated on surgical pathology

SECONDARY OUTCOMES:
Ki-67 concordance | 18 months
  To evaluate the concordance rate of Ki67-based tumor grade between endoscopic ultrasound biopsy samples and surgical specimens.
DAXX/ATRX concordance | 18 months
  To evaluate the concordance rate of DAXX/ATRX expression between endoscopic ultrasound biopsy samples and surgical specimens
Ki-67-tumor aggressiveness association | 18 months
  To assess the association between preoperative Ki67-based grade 2/3 on endoscopic ultrasound samples and pathological features indicative of tumor aggressiveness evaluated on surgical pathology
Preoperative prognosis assessment | 60 months
  To evaluate the association between DAXX/ATRX expression on endoscopic ultrasound biopsy samples, Ki67-based grade 2/3 on endoscopic ultrasound biopsy samples, and tumor size on endoscopic ultrasound and progression-free survival and relapse-free survival.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Verona, Verona, Italy